CLINICAL TRIAL: NCT06363097
Title: The Effect of Dietary Sodium Intake on Ambulatory Blood Pressure Levels According to Urinary Uromodulin Levels in Patients With Chronic Kidney Disease
Brief Title: Urinary Uromodulin, Dietary Sodium Intake and Ambulatory Blood Pressure in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: ΔΔ5032
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: CKD; Uromodulin; sodium intake
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low uromodulin group: Patients with urinary uromodulin levels below median.
- High uromodulin group: Patients with urinary uromodulin levels above median.

SUMMARY:
In chronic kidney disease (CKD), hypertension is characterized by the phenomenon of sodium-sensitivity, i.e., the disproportionate increase in blood pressure (BP) due to an increase in dietary sodium consumption to maintain homeostasis through urinary sodium excretion. Impaired renal circulation, blunt suppression of renin-angiotensin-aldosterone system, sympathetic nervous system overactivity, paradoxically reduced levels of atrial natriuretic peptide and hyperinsulinemia represent the main pathophysiologic mechanisms. Accumulated evidence has suggested that uromodulin plays a central role in the development of sodium-sensitive hypertension. Uromodulin is a kidney-specific glycoprotein which is exclusively produced by the epithelial cells lining the thick ascending limb and early distal convoluted tubule. It is currently recognized as a multifaceted player in kidney physiology and disease, with discrete roles for intracellular, urinary, interstitial and serum uromodulin. Among these, urinary uromodulin modulates renal sodium handling through regulating tubular transporters that reabsorb sodium and are targeted by diuretics, i.e., the loop diuretic-sensitive Na+-K+-2Cl- cotransporter type 2 (NKCC2) and the thiazide-sensitive Na+/Cl- cotransporter (NCC). Given these roles, the contribution of uromodulin to sodium-sensitive hypertension has been proposed. In preclinical models, uromodulin deficiency causes decreased BP that is resistant to dietary salt, while uromodulin overexpression causes hypertension due to increased tubular sodium reabsorption that is responsive to furosemide. Genetic human studies have identified robust associations of specific UMOD gene variants with sodium sensitivity and incident hypertension risk, while comprehensive Mendelian randomization studies have affirmed these associations by highlighting the causal relationship between UMOD variants, urinary uromodulin levels and hypertension. Furthermore, clinical studies in both healthy individuals and hypertensive patients have indicated a link between sodium sensitivity and uromodulin, directly affecting mean BP levels and BP response to salt intake. With regards to CKD population, solid data on the link of uromodulin with sodium sensitivity are currently missing from the literature. There is only a pediatric study in the setting of CKD (stages 2-3), which failed to show an association between urinary uromodulin levels indexed to urinary creatinine (UMOD/uCr) and either 24-hour or office BP; however, this study has several limitations, and its results should be interpreted with caution. To best of our knowledge, there is no study up to date investigating the effect of dietary sodium intake on 24-hour ambulatory blood pressure depending on urinary uromodulin levels in adult CKD patients.

DETAILED DESCRIPTION:
This is a cross-sectional study performed in the 1st Department of Nephrology, Hippokration Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece. For the purposes of this study, adult (aged ≥18 years) CKD patients (defined based on the KDIGO criteria) fulfilling the inclusion and exclusion criteria were invited to participate. All included patients signed a written informed consent form prior to study enrollment. The study protocol was approved by the Ethics Committee of the School of Medicine, Aristotle University of Thessaloniki and the and the Institutional Review Board of Hippokration Hospital, Thessaloniki, Greece. All procedures and evaluations are performed according to the Declaration of Helsinki 2013 Amendment and directives of the General Data Protection Regulation (GDPR).

Baseline evaluation includes the recording of demographics, anthropometric characteristics, CKD cause, comorbidities, concomitant medications, as well as a detailed physical examination and venous blood sampling for routine laboratory tests. Study participants are advised to refrain from food, caffeine, alcohol, or tobacco for 12 h and receive any standard medication before their morning appointment in the research laboratory to perform the assessments described below. Office BP measurements are performed thrice after 5-10 min of rest, in the sitting position, at the level of the brachial artery, with a validated oscillometric device [Omron M3 Intellisense (Omron Healthcare, Kyoto, Japan)] using a cuff of appropriate size, according to current guidelines. Afterwards, evaluation of patient's hydration status will be performed with lung ultrasound [GE VScan (GE Healthcare, Horten, Norway)] through quantification of US-B lines. The Mini-Mental State Exam (MMSE) is used for the assessment of cognitive function; sleep quality is evaluated by the Pittsburg Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS), while the severity of nocturia is also recorded. Following that, patients will undergo a 24-hour ambulatory BP monitoring (ABPM) with ABPMpro (SOMNOmedics, Randersacker, Germany) with an appropriately sized cuff. The device will take measurements every 20 minutes between 07:00 and 23:00 (daytime period) and every 30 minutes between 23:00 and 07:00 (nighttime period). Simultaneously, patients will perform a 24-hour urine collection, divided in two distinct periods (daytime and nighttime) with the use of two different containers matching the corresponding ABPM periods.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. CKD defined based on the KDIGO criteria
3. Provision of informed written consent

Exclusion Criteria:

1. Kidney transplantation or end-stage kidney disease (ESKD) under hemodialysis or peritoneal dialysis
2. Chronic atrial fibrillation or other diagnosed arrhythmia intervening with a proper 24-hour ABPM recording
3. Inability to reliably complete the study questionnaires
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients with CKD across all consecutive pre-dialysis stages.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Effect of urinary uromodulin levels on the relationship between 24-hour urinary sodium excretion and 24-hour ambulatory systolic blood pressure. | Baseline
  In patients with high and low urinary uromodulin excretion, investigation of the relationship of 24-hour urinary sodium excretion with 24-hour ambulatory systolic blood pressure.
Effect of urinary uromodulin levels on the relationship between 24-hour urinary sodium excretion and 24-hour ambulatory diastolic blood pressure. | Baseline
  In patients with high and low urinary uromodulin excretion, investigation of the relationship of 24-hour urinary sodium excretion with 24-hour ambulatory diastolic blood pressure.

SECONDARY OUTCOMES:
Effect of urinary uromodulin levels on the relationship between nighttime/daytime ratio of urinary sodium excretion and 24-hour ambulatory systolic blood pressure. | Baseline
  In patients with high and low urinary uromodulin excretion, investigation of the relationship between nighttime/daytime ratio of urinary sodium excretion and 24-hour ambulatory systolic blood pressure.
Effect of urinary uromodulin levels on the relationship between nighttime/daytime ratio of urinary sodium excretion and 24-hour ambulatory diastolic blood pressure. | Baseline
  In patients with high and low urinary uromodulin excretion, investigation of the relationship between nighttime/daytime ratio of urinary sodium excretion and 24-hour ambulatory diastolic blood pressure.
Effect of urinary uromodulin levels on the relationship between urinary sodium-to-potassium (Na+/K+) ratio and 24-hour ambulatory systolic blood pressure. | Baseline
  In patients with high and low urinary uromodulin excretion, investigation of the relationship between urinary sodium-to-potassium (Na+/K+) ratio and 24-hour ambulatory systolic blood pressure.
Effect of urinary uromodulin levels on the relationship between urinary sodium-to-potassium (Na+/K+) ratio and 24-hour ambulatory diastolic blood pressure. | Baseline
  In patients with high and low urinary uromodulin excretion, investigation of the relationship between urinary sodium-to-potassium (Na+/K+) ratio and 24-hour ambulatory diastolic blood pressure.
The difference in 24-hour ambulatory brachial SBP/DBP between patients with high and low urinary uromodulin excretion. | Baseline
The difference in 24-hour ambulatory brachial SBP/DBP standard deviation (SD) between patients with high and low urinary uromodulin excretion. | Baseline
The difference in 24-hour ambulatory brachial SBP/DBP weighted SD (wSD) between patients with high and low urinary uromodulin excretion. | Baseline
The difference in 24-hour ambulatory brachial SBP/DBP coefficient of variation (CV) between patients with high and low urinary uromodulin excretion. | Baseline
The difference in 24-hour ambulatory brachial SBP/DBP average real variability (ARV) between patients with high and low urinary uromodulin excretion. | Baseline
Effect of 24-hour urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP standard deviation (SD). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of 24-hour urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP weighted SD (wSD). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of 24-hour urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP coefficient of variation (CV). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of 24-hour urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP average real variability (ARV). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of nighttime/daytime ratio of urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP standard deviation (SD). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of nighttime/daytime ratio of urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP weighted SD (wSD). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of nighttime/daytime ratio of urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP coefficient of variation (CV). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of nighttime/daytime ratio of urinary sodium excretion on 24-hour ambulatory brachial SBP/DBP average real variability (ARV). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of urinary sodium-to-potassium (Na+/K+) ratio on 24-hour ambulatory brachial SBP/DBP standard deviation (SD). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of urinary sodium-to-potassium (Na+/K+) ratio on 24-hour ambulatory brachial SBP/DBP weighted SD (wSD). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of urinary sodium-to-potassium (Na+/K+) ratio on 24-hour ambulatory brachial SBP/DBP coefficient of variation (CV). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of urinary sodium-to-potassium (Na+/K+) ratio on 24-hour ambulatory brachial SBP/DBP average real variability (ARV). | Baseline
  (This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the ABPMpro device).
Effect of 24-hour urinary sodium excretion on hydration status (US-B lines). | Baseline
  (The hydration status will be assessed through quantification of US-B lines using GE VScan lung ultrasound device).
Effect of nighttime/daytime ratio of urinary sodium excretion on hydration status (US-B lines). | Baseline
  (The hydration status will be assessed through quantification of US-B lines using GE VScan lung ultrasound device).
Effect of urinary sodium-to-potassium (Na+/K+) ratio on hydration status (US-B lines). | Baseline
  (The hydration status will be assessed through quantification of US-B lines using GE VScan lung ultrasound device).
Effect of 24-hour urinary sodium excretion on MMSE score. | Baseline
Effect of nighttime/daytime ratio of urinary sodium excretion on MMSE score. | Baseline
Effect of urinary sodium-to-potassium (Na+/K+) ratio on MMSE score. | Baseline
Effect of 24-hour urinary sodium excretion on PSQI score. | Baseline
Effect of nighttime/daytime ratio of urinary sodium excretion on PSQI score. | Baseline
Effect of urinary sodium-to-potassium (Na+/K+) ratio on PSQI score. | Baseline
Effect of 24-hour urinary sodium excretion on ESS score. | Baseline
Effect of nighttime/daytime ratio of urinary sodium excretion on ESS score. | Baseline
Effect of urinary sodium-to-potassium (Na+/K+) ratio on ESS score. | Baseline
Effect of 24-hour urinary sodium excretion on nocturnal urinations. | Baseline
Effect of nighttime/daytime ratio of urinary sodium excretion on nocturnal urinations. | Baseline
Effect of urinary sodium-to-potassium (Na+/K+) ratio on nocturnal urinations. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Nephrology, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karagiannidis AG, Theodorakopoulou MP, Pella E, Sarafidis PA, Ortiz A. Uromodulin biology. Nephrol Dial Transplant. 2024 Jun 28;39(7):1073-1087. doi: 10.1093/ndt/gfae008. PMID 38211973
- [Background] Padmanabhan S, Melander O, Johnson T, Di Blasio AM, Lee WK, Gentilini D, Hastie CE, Menni C, Monti MC, Delles C, Laing S, Corso B, Navis G, Kwakernaak AJ, van der Harst P, Bochud M, Maillard M, Burnier M, Hedner T, Kjeldsen S, Wahlstrand B, Sjogren M, Fava C, Montagnana M, Danese E, Torffvit O, Hedblad B, Snieder H, Connell JM, Brown M, Samani NJ, Farrall M, Cesana G, Mancia G, Signorini S, Grassi G, Eyheramendy S, Wichmann HE, Laan M, Strachan DP, Sever P, Shields DC, Stanton A, Vollenweider P, Teumer A, Volzke H, Rettig R, Newton-Cheh C, Arora P, Zhang F, Soranzo N, Spector TD, Lucas G, Kathiresan S, Siscovick DS, Luan J, Loos RJ, Wareham NJ, Penninx BW, Nolte IM, McBride M, Miller WH, Nicklin SA, Baker AH, Graham D, McDonald RA, Pell JP, Sattar N, Welsh P; Global BPgen Consortium; Munroe P, Caulfield MJ, Zanchetti A, Dominiczak AF. Genome-wide association study of blood pressure extremes identifies variant near UMOD associated with hypertension. PLoS Genet. 2010 Oct 28;6(10):e1001177. doi: 10.1371/journal.pgen.1001177. PMID 21082022
- [Background] Trudu M, Janas S, Lanzani C, Debaix H, Schaeffer C, Ikehata M, Citterio L, Demaretz S, Trevisani F, Ristagno G, Glaudemans B, Laghmani K, Dell'Antonio G; SKIPOGH team; Loffing J, Rastaldi MP, Manunta P, Devuyst O, Rampoldi L. Common noncoding UMOD gene variants induce salt-sensitive hypertension and kidney damage by increasing uromodulin expression. Nat Med. 2013 Dec;19(12):1655-60. doi: 10.1038/nm.3384. Epub 2013 Nov 3. PMID 24185693
- [Background] Ponte B, Sadler MC, Olinger E, Vollenweider P, Bochud M, Padmanabhan S, Hayward C, Kutalik Z, Devuyst O. Mendelian randomization to assess causality between uromodulin, blood pressure and chronic kidney disease. Kidney Int. 2021 Dec;100(6):1282-1291. doi: 10.1016/j.kint.2021.08.032. Epub 2021 Oct 9. PMID 34634361
- [Background] Ponte B, Pruijm M, Ackermann D, Olinger E, Youhanna S, Vogt B, Burnier M, Pechere-Bertschi A, Bochud M, Devuyst O. Uromodulin, Salt, and 24-Hour Blood Pressure in the General Population. Clin J Am Soc Nephrol. 2021 May 8;16(5):787-789. doi: 10.2215/CJN.11230720. Epub 2021 Jan 21. No abstract available. PMID 33478975
- [Background] Torffvit O, Melander O, Hulten UL. Urinary excretion rate of Tamm-Horsfall protein is related to salt intake in humans. Nephron Physiol. 2004;97(1):p31-6. doi: 10.1159/000077600. PMID 15153749
- [Background] Bakhoum CY, Anderson CAM, Juraschek SP, Rebholz CM, Appel LJ, Miller ER, Parikh CR, Obeid W, Rifkin DE, Ix JH, Garimella PS. The Relationship Between Urine Uromodulin and Blood Pressure Changes: The DASH-Sodium Trial. Am J Hypertens. 2021 Mar 11;34(2):154-156. doi: 10.1093/ajh/hpaa140. PMID 32856709
- [Background] Bakhoum CY, Matheson MB, Greenberg JH, Furth SL, Ix JH, Garimella PS. Urine Uromodulin Is Not Associated With Blood Pressure in the Chronic Kidney Disease in Children Cohort. Hypertension. 2022 Oct;79(10):2298-2304. doi: 10.1161/HYPERTENSIONAHA.122.19566. Epub 2022 Aug 3. PMID 35920156
- [Background] McCallum L, Brooksbank K, McConnachie A, Aman A, Lip S, Dawson J, MacIntyre IM, MacDonald TM, Webb DJ, Padmanabhan S. Rationale and Design of the Genotype-Blinded Trial of Torasemide for the Treatment of Hypertension (BHF UMOD). Am J Hypertens. 2021 Feb 18;34(1):92-99. doi: 10.1093/ajh/hpaa166. PMID 33084880